CLINICAL TRIAL: NCT00921687
Title: Chronic Kidney Disease Guideline Adherence - a Cluster Randomized Controlled Quality Improvement Study
Brief Title: Chronic Kidney Disease (CKD) Guideline Adherence - A Quality Improvement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Drawz, Senior Instructor, Louis Stokes VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LSCVAMCCKD1
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifactorial intervention (Experimental): The multifactorial intervention will consist of a CKD lecture, the CKD reference card, academic detailing, and access to the CKD registry.
  Interventions: Behavioral: Multifactorial intervention
- Education only (Active Comparator): Providers in the education only arm will receive a CKD lecture and be given a CKD reference card.
  Interventions: Behavioral: Education only

INTERVENTIONS:
Behavioral: Education only — The education will consist of a lecture and distribution of a CKD reference card.
  Arms: Education only
Behavioral: Multifactorial intervention — Providers in the intervention group will receive a lecture on CKD, a CKD reference card, academic detailing (residents only), and access to the CKD registry.
  Arms: Multifactorial intervention

SUMMARY:
Chronic kidney disease (CKD) is defined as kidney damage for greater than 3 months or a glomerular filtration rate less than 60 mL/min per 1.73m2 for greater than 3 months. Patients with CKD are at high risk for development of cardiovascular disease and metabolic complications. Guidelines for the care of patients with CKD have been developed by the National Kidney Foundation. Despite the wide availability of these guidelines, adherence is low. The goal of the current study is to evaluate whether a multifactorial intervention, including a CKD registry, will improve CKD guideline adherence. The hypothesis is that providers exposed to a multifactorial clinical intervention including education, academic detailing, and a CKD registry will be more likely to adhere to CKD guidelines than those only exposed to education.

ELIGIBILITY:
Providers:

Inclusion Criteria:

* All primary care providers at the Wade Park Veterans Affairs Medical Center (VAMC) will be eligible for the study

Patients:

Inclusion Criteria:

* Receive primary care from a provider at the Wade Park VAMC
* Have:

  * CKD as defined by an estimated glomerular filtration rate (eGFR) less than 60 on two separate occasions 90 to 730 days apart,
  * diabetes, OR
  * hypertension

Exclusion Criteria:

* End-stage renal disease
* Renal transplant recipients
* Less than 18 years of age on July 1, 2009
* No primary care visit between Jan 1, 2008 and July 1, 2009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Drawz, MD, MHS, MS, Principal Investigator — Louis Stokes VA Medical Center
Locations (1):
- Louis Stokes Cleveland Veterans Affairs Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Hoy T, Fisher M, Barber B, Borker R, Stolshek B, Goodman W. Adherence to K/DOQI practice guidelines for bone metabolism and disease. Am J Manag Care. 2007 Nov;13(11):620-5. PMID 17988187
- [Background] Philipneri MD, Rocca Rey LA, Schnitzler MA, Abbott KC, Brennan DC, Takemoto SK, Buchanan PM, Burroughs TE, Willoughby LM, Lentine KL. Delivery patterns of recommended chronic kidney disease care in clinical practice: administrative claims-based analysis and systematic literature review. Clin Exp Nephrol. 2008 Feb;12(1):41-52. doi: 10.1007/s10157-007-0016-3. Epub 2008 Jan 5. PMID 18175059
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Derived] Drawz PE, Miller RT, Singh S, Watts B, Kern E. Impact of a chronic kidney disease registry and provider education on guideline adherence--a cluster randomized controlled trial. BMC Med Inform Decis Mak. 2012 Jul 5;12:62. doi: 10.1186/1472-6947-12-62. PMID 22765882
- See also: abstract - BMC Medical Informatics and Decision Making — http://www.biomedcentral.com/1472-6947/12/62/abstract

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Providers in the control group received education only (CKD lecture and a CKD reference card).
- Intervention: The multifactorial intervention consisted of a CKD lecture, the CKD reference card, academic detailing, and access to the CKD registry.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 418 (eligible patients seen in clinic between 1/1/09 and 1/1/10) | 363
Completed | 418 | 363
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Clinic: Providers in the control group received education only (chronic kidney disease (CKD) lecture and a CKD reference card).
- Intervention Clinic: The multifactorial intervention consisted of a CKD lecture, the CKD reference card, academic detailing, and access to the CKD registry.
- Total: Total of all reporting groups
Arm/Group | Control Clinic | Intervention Clinic | Total
Number analyzed (Participants) | 418 | 363 | 781
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (10.3) | 71 (10.7) | 71 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 401 | 343 | 744
Diabetes [Number; unit: participants]
  Yes | 210 | 163 | 373
  No | 208 | 200 | 408
Hypertension [Number; unit: participants]
  Yes | 389 | 352 | 741
  No | 29 | 11 | 40
Stage of chronic kidney disease [Number; unit: participants] — Stage III - estimated glomerular filtration rate (eGFR) <60 and >=30 Stage IV - eGFR <30 and >=15 Stage V - eGFR <15 Stage V is the worst clinical stage (lower eGFR indicates worse kidney function).
  participants
    Stage III | 383 | 325 | 708
    Stage IV | 32 | 36 | 68
    Stage V | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: PTH (Parathyroid Hormone) Adherence
Description: Probability for having a PTH measured during the study period comparing intervention vs control clinic during the study period as estimated by Generalized Estimating Equation (determines probability, not proportion). Participants assigned 1 if PTH was measured and 0 if PTH was not measured during the study period.
Time Frame: One year
Measure: Number; unit: probability of having a PTH measured
Arm/Group | Control Clinic | Intervention Clinic
Number analyzed (Participants) | 418 | 363
probability of having a PTH measured | 0.23 | 0.28
Statistical Analysis 1: Comparison: Control Clinic vs Intervention Clinic; Test type: Superiority or Other; p = 0.04, Generalized Estimating Equation; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.01 to 2.30] — Intervention clinic (vs control clinic)

2. Secondary Outcome: Last Clinic BP <130/80 mmHg
Description: Probability of last Clinic BP <130/80 mmHg Comparing Intervention vs Control Clinic During the Study Period as estimated using Generalized Estimating Equation.
Time Frame: One year
Measure: Number (95% Confidence Interval); unit: probability of controlled clinic BP
Arm/Group | Control Clinic | Intervention Clinic
Number analyzed (Participants) | 418 | 363
probability of controlled clinic BP | 0.41 [0.36 to 0.46] | 0.44 [0.39 to 0.49]
Statistical Analysis 1: Comparison: Control Clinic vs Intervention Clinic; Test type: Superiority or Other; p = 0.44, Generalized Estimating Equation; Odds Ratio (OR) = 1.12, 95% CI [0.84 to 1.49] — Intervention clinic (vs control clinic)

ADVERSE EVENTS:
Arm/Group | Control Clinic | Intervention Clinic
Serious Adverse Events (participants affected / at risk) | 0/418 | 0/363
Other Adverse Events (participants affected / at risk) | 0/418 | 0/363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes